CLINICAL TRIAL: NCT03815513
Title: Non-invasive Evaluation of Cerebrovascular Reactivity in Spontaneous Intracerebral Hemorrhage
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201811003RINB
Record Dates: First submitted 2019-01-17; First posted 2019-01-24 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2018-12

CONDITIONS: Intracerebral Hemorrhage
Keywords: Intracerebral hemorrhage; MRI; human
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Intervention Model Description: Both patient with intracerebral hemorrhage and healthy control will receive brain MRI with Dipyridamole stimulation for cerebrovascular reactivity measurement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cases (Experimental): Patient with spontaneous intracerebral hemorrhage
  Interventions: Other: brain MRI
- controls (Experimental): Healthy control without history of symptomatic cerebrovascular diseases
  Interventions: Other: brain MRI

INTERVENTIONS:
Other: brain MRI — both case and control groups received brain MRI to evaluate cerebrovascular reactivity

SUMMARY:
Spontaneous intracerebral hemorrhage (ICH) remains a significant cause of morbidity and mortality around the globe. The most common etiology of nontraumatic spontaneous ICH is hypertensive arteriopathy (HA), while cerebral amyloid angiopathy (CAA) is the most prevalent cause of spontaneous lobar ICH in the elderly. Both HA and CAA belong to the family of cerebral small vessel disease (cSVD). cSVD involves pathological processes that affect the arteries, arterioles, capillaries, and veins on the surface and beneath the brain. The resultant changes of cSVD in the brain vasculatures can be detected with neuroimaging, includes cerebral microbleeds, white matter hyperintensities, lacunes, dilated perivascular spaces, and brain atrophy.

Investigators of this study have probe into various imaging markers in patients with cSVD. Investigators found that the lacune and cerebral microbleeds location was related to distinct underlying etiology of cSVD. Further, investigators utilized amyloid PET study to directly quantified the cerebral amyloid burden, and demonstrated the correlation between amyloid deposition and deep/superficial microbleeds ratio. The association between cerebellum microbleeds, which is a novel marker for cSVD, and the underlying pathology in patient with spontaneous ICH has been investigated. Investigators also summarized and published the current research of different cSVD imaging markers and its implication on patient care.

Cerebrovascular reactivity (CVR) represents the phenomenon that cerebral vessels dilate or constrict in response to stimuli, which provides insights into the vascular reserve information. The vascular reserve parameter is complementary to steady-state vascular index, such as cerebral perfusion or other neuroimaging markers. Measurement of CVR using advanced MR techniques is an emerging technique with multiple potential clinical utilities, and impaired autoregulation may contribute to the pathogenesis of cSVD. Recently, diminished CVR under visual stimuli has been linked to vascular amyloid deposits and related vascular dysfunction. Clarifying the mechanism of cSVD-related brain injury would be an important step towards identifying candidate treatment approaches.

The goal of this study is to understand the features of CVR in patients with cSVD-related spontaneous ICH, for the purpose of establishing new biomarkers in cSVD diagnosis and understanding the underlying pathophysiology.

ELIGIBILITY:
Inclusion Criteria:

* age between 20-90 years-old
* patient with spontaneous intracerebral hemorrhage or healthy control
* consciousness clear
* willing to receive brain MRI

Exclusion Criteria:

* renal failure or Creatinine > 2mg/dl
* coagulopathy or hepatic insufficiency
* unstable vital sign under inotropic agents
* allergy to Dipyridamole
* pregnancy
* asthma history
* metal implant or cardiac pacemaker

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01-21 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Intracerebral hemorrhage recurrence | The patients will be follow up in the outpatient clinic for 2 years.
  Symptomatic intracerebral hemorrhage recurrence during follow-up
Ischemic stroke recurrence | The patients will be follow up in the outpatient clinic for 2 years.
  Symptomatic ischemic stroke recurrence during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tsai HH, Pasi M, Tsai LK, Chen YF, Lee BC, Tang SC, Fotiadis P, Huang CY, Yen RF, Gurol ME, Jeng JS. Distribution of Lacunar Infarcts in Asians With Intracerebral Hemorrhage: A Magnetic Resonance Imaging and Amyloid Positron Emission Tomography Study. Stroke. 2018 Jun;49(6):1515-1517. doi: 10.1161/STROKEAHA.118.021539. Epub 2018 Apr 25. PMID 29695464
- [Background] Tsai HH, Tsai LK, Chen YF, Tang SC, Lee BC, Yen RF, Jeng JS. Correlation of Cerebral Microbleed Distribution to Amyloid Burden in Patients with Primary Intracerebral Hemorrhage. Sci Rep. 2017 Mar 17;7:44715. doi: 10.1038/srep44715. PMID 28303922
- [Background] Dumas A, Dierksen GA, Gurol ME, Halpin A, Martinez-Ramirez S, Schwab K, Rosand J, Viswanathan A, Salat DH, Polimeni JR, Greenberg SM. Functional magnetic resonance imaging detection of vascular reactivity in cerebral amyloid angiopathy. Ann Neurol. 2012 Jul;72(1):76-81. doi: 10.1002/ana.23566. PMID 22829269
- [Background] Fisher M, Vasilevko V, Passos GF, Ventura C, Quiring D, Cribbs DH. Therapeutic modulation of cerebral microhemorrhage in a mouse model of cerebral amyloid angiopathy. Stroke. 2011 Nov;42(11):3300-3. doi: 10.1161/STROKEAHA.111.626655. Epub 2011 Sep 8. PMID 21903962